CLINICAL TRIAL: NCT05393453
Title: The Investigate Outcomes and Prognostic Factors of Patients With Acute-on-chronic Liver Failure
Brief Title: Prognosis of Patients With Acute-on-chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: Xiangya ACLF project
Record Dates: First submitted 2022-05-14; First posted 2022-05-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood includes blood cells and serum, urine and fecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with acute on chronic liver failure: All subjects will receive the currently routine treatment of liver failure and corresponding etiological treatment if needed. The researchers will collect various clinical examination results of the subjects in the process of diagnosis and treatment, including but not limited to blood routine, biochemistry, coagulation function, liver imaging, therapeutic drugs, etc. Complications and prognosis of patients will be recorded. Blood samples, urine and stool samples of all subjects will be collected after enrollment and stored for probably testing in the future. This study has no additional intervention and treatment for subjects.

SUMMARY:
Patients with Acute on Chronic Liver Failure (ACLF) have high short-term mortality. The use of a severity score could define the patient's prognosis. This study mainly prospectively analyze the clinical data of patients with chronic liver disease related acute liver failure admitted to the department of infectious diseases, Xiangya Hospital of Central South University, to analyze the prognosis of patients with chronic liver disease related acute on-chronic liver failure in Central South China. No additional interventions other than routine treatment will be added.

DETAILED DESCRIPTION:
Patients with Acute on Chronic Liver Failure (ACLF) have high short-term mortality. The use of a severity score could define the patient's prognosis and would help determine in whom the treatment is effective. This study mainly prospectively analyze the clinical data of patients with chronic liver disease related acute liver failure admitted to the department of infectious diseases, Xiangya Hospital of Central South University, to analyze the short-time and relatively long-term prognosis of patients with chronic liver disease related acute on-chronic liver failure. This is an observational study. All subjects will receive the currently recognized routine treatment of liver failure and corresponding etiological treatment if needed. The researchers will collect various clinical examination indexes of the subjects in the process of diagnosis and treatment, including but not limited to blood routine, biochemistry, coagulation function, liver imaging, therapeutic drugs, etc. Complications and prognosis of patients will be recorded. Blood samples, urine and stool samples of all subjects will be taken after enrollment and stored for probably testing in the future. This study has no additional intervention and treatment for subjects. All subjects will sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* patients with evidence of chronic liver disease patients with liver failure

Exclusion Criteria:

* Patients who do not have chronic liver disease Patients who have hepatocellular carcinoma Patients who admitted for extrahepatic manifestations Patients who have HIV infection Patients who admitted for symptomatic control of chronic liver disease, other than acute deterioration of liver function

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with any cause of chronic liver disease who underwent acute liver dysfunction meets the criteria of ACLF of APASL.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Non-liver transplant mortality | 15 days
  short time mortality
Non-liver transplant mortality | 30 days
  short time mortality
Non-liver transplant mortality | 90 days
  short time mortality
Non-liver transplant mortality | 12 months
  long time mortality
Non-liver transplant mortality | 36 months
  long time mortality

SECONDARY OUTCOMES:
Liver transplantation rate | 1 month
  mortality of all patients including those receiving liver transplantation
Liver transplantation rate | 6 months
  mortality of all patients including those receiving liver transplantation
Liver transplantation rate | 12 months
  mortality of all patients including those receiving liver transplantation
Model for disease severity | 1 month
  MELD score will be calculated and reported
Model for disease severity | 6 months
  MELD score will be calculated and reported
Model for disease severity | 12 months
  MELD score will be calculated and reported

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided